CLINICAL TRIAL: NCT03777241
Title: Disruptive bEhavior manageMEnt ANd Prevention in Hospitalized Patients Using a behaviORal Intervention Team: Study Protocol for a Pragmatic, Cluster, Cross-over Design
Brief Title: Disruptive bEhavior manageMEnt ANd Prevention in Hospitalized Patients Using a behaviORal Intervention Team
Acronym: DEMEANOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Ruth Kleinpell, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 182229
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Behavioral Problem
MeSH Terms: conditions — Problem Behavior | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention Team (Active Comparator): The participants in this arm will receive the Behavioral Intervention Team.
  Interventions: Behavioral: Behavioral Intervention Team
- Standard of Care (Active Comparator): The participants in this arm will receive the standard of care.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Behavioral Intervention Team — Multidisciplinary team to assist with actively identifying and managing mental illness and substance abuse disorders at their earliest possible time during hospitalization.
  Arms: Behavioral Intervention Team
Behavioral: Standard of care — Participants in this group will receive standard of care.
  Arms: Standard of Care

SUMMARY:
The purpose of the proposed study is to evaluate the impact of a behavioral intervention team (BIT) on 2 adult units: a general medical (8N); a cardiac/medical stepdown (8S) at Vanderbilt University Medical Center (VUMC) with a higher proportion of patients with behavioral health comorbidities.

DETAILED DESCRIPTION:
The BIT will provide a proactive psychiatric team that will screen all patients on admission, provide consultation to those meeting established criteria, and recommend interventions to the primary care team for consideration. BIT will also serve to model therapeutics tactics in communication and goal setting to the clinical staff.

Research Questions for the proposed study:

Considering that behavioral health co-morbidity is common among hospitalized medical inpatients and is associated with higher costs of care and staff dissatisfaction, we will ascertain whether the addition of dedicated, trained behavioral intervention team, compared to nursing staff training on trauma informed care and de-escalation techniques provides:

1. meaningful, measureable improvement in the prevention and management of disruptive behavior in the healthcare setting at VUMC, and
2. Improvement in staff perceptions of their ability to manage patients exhibiting disruptive, threatening or acting out behavior

Specifically, using a pragmatic, cluster cross-over trial design where the BIT crosses between 8N and 8S, we will test the hypothesis that presence of the BIT results in:

1. Improvement in the prevention and management of patients exhibiting disruptive, threatening or acting out behavior
2. Improvement in staff perceptions of their ability to manage patients exhibiting disruptive, threatening or acting out behavior

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to two adult medical surgical units (8N/8S) at Vanderbilt University Medical Center during the study period.
* All clinical nurses and staff on 8N/8S employed during the study period.

Exclusion Criteria:

* Patients admitted to the floor before the BIT team has begun the crossover period on the unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3800 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Percent of violence control measures utilized | 6 months
  By extracting medications, restraints, and sitters ordered from the electronic health records
Percent of patient injurious behaviors reported | 6 months
  By extracting reports of biting, kicking, throwing, etc. from the electronic medical record
Percent change in nurse comfort and confidence in their ability to manage patients exhibiting disruptive, threatening or acting out behavior | 1 year
  By administering surveys to participants

SECONDARY OUTCOMES:
Rate of unit nursing staff retention | 1 year
  By extracting rates from internal human resources records
Patient length of stay | 6 months
  By extracting data from the electronic health record

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Kleinpell, PhD, RN, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data be available (including data dictionaries) will be shared, particularly individual participant data that underlie the results reported after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Proposals should be directed to the PI via the Learning Healthcare System platform secondary data use application
URL: https://redcap.vanderbilt.edu/surveys/?s=CR8TNYXKWX

REFERENCES:
- [Derived] Hasselblad M, Morrison J, Kleinpell R, Buie R, Ariosto D, Hardiman E, Osborn SW, Nwosu SK, Lindsell C. Promoting patient and nurse safety: testing a behavioural health intervention in a learning healthcare system: results of the DEMEANOR pragmatic, cluster, cross-over trial. BMJ Open Qual. 2022 Feb;11(1):e001315. doi: 10.1136/bmjoq-2020-001315. PMID 35131740
- [Derived] Morrison J, Hasselblad M, Kleinpell R, Buie R, Ariosto D, Hardiman E, Osborn SW, Lindsell CJ; Vanderbilt Learning Healthcare System Investigators, Vanderbilt University. The Disruptive bEhavior manageMEnt ANd prevention in hospitalized patients using a behaviORal intervention team (DEMEANOR) study protocol: a pragmatic, cluster, crossover trial. Trials. 2020 May 24;21(1):417. doi: 10.1186/s13063-020-04278-2. PMID 32448331